CLINICAL TRIAL: NCT03467217
Title: Losartan for the Treatment of Pediatric NAFLD (STOP-NAFLD): A Phase 2, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Losartan for the Treatment of Pediatric NAFLD
Acronym: STOP-NAFLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial stopped for futility
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9 STOP-NAFLD; U01DK061730 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease
Keywords: Losartan; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators, clinical staff, and data monitoring committee will not have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan potassium capsule (Active Comparator): Dose will be one 50 mg capsule of losartan per day for one week and then increased to two capsules of 50 mg of losartan per day (100 mg total) for 23 weeks patients with baseline weight ≥ 70 kg to <150 kg.
  Interventions: Drug: Losartan potassium
- Placebo losartan capsule (Placebo Comparator): Dose will be one 50 mg capsule of placebo losartan per day for one week and then increased to two capsules of 50 mg of placebo losartan per day (100 mg total) for 23 weeks for patients with baseline weight ≥ 70 kg to <150 kg.
  Interventions: Drug: Placebo losartan capsule

INTERVENTIONS:
Drug: Losartan potassium — Losartan potassium is an angiotensin II receptor blocker acting on the AT 1 receptor subtype
  Other Names: losartan, Cozaar,
  Arms: Losartan potassium capsule
Drug: Placebo losartan capsule — Matching placebo losartan oral capsule
  Arms: Placebo losartan capsule

SUMMARY:
A multicenter, randomized, double masked, placebo-controlled, parallel treatment groups phase 2 trial of losartan for pediatric nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Children ages 8-17 years weighing between 70 -149 kilograms will be enrolled and treated with losartan (100 mg orally once per day) or matching placebo for 24 weeks. The hypothesis is that losartan will improve serum alanine aminotransferase (ALT) in children with pediatric NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years at initial screening interview
* Histological evidence of NAFLD with or without fibrosis and a NAFLD activity score (NAS) of ≥3, on a liver biopsy obtained no more than 730 days prior to enrollment.
* Serum ALT at screening ≥ 50 IU/L

Exclusion Criteria:

* Body weight less than 70 kg or greater than 150 kg at screening
* Significant alcohol consumption or inability to reliably quantify alcohol intake
* Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, other known hepatotoxins) for more than 2 consecutive weeks in the past year prior to randomization
* New treatment with vitamin E or metformin started in the past 90 days or plans to alter the dose or stop over the next the 24 weeks. A stable dose is acceptable.
* Prior or planned bariatric surgery
* Uncontrolled diabetes (HbA1c 9.5% or higher)
* Presence of cirrhosis on liver biopsy
* History of hypotension or history of orthostatic hypotension
* Stage 2 Hypertension or >140 systolic or >90 diastolic at screening
* Current treatment with any antihypertensive medications including all angiotensin converting enzyme (ACE) inhibitors or aliskiren
* Current treatment with potassium supplements or any drug known to increase potassium
* Current daily use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Current treatment with lithium
* Platelet counts below 100,000 /mm3
* Clinical evidence of hepatic decompensation (serum albumin < 3.2 g/dL, international normalized ratio (INR) >1.3, direct bilirubin >1.3 mg/dL, history of esophageal varices, ascites, or hepatic encephalopathy)
* Evidence of chronic liver disease other than NAFLD:

  * Biopsy consistent with histological evidence of autoimmune hepatitis
  * Serum hepatitis B surface antigen (HBsAg) positive.
  * Serum hepatitis C antibody (anti-HCV) positive.
  * Iron/total iron binding capacity (TIBC) ratio (transferrin saturation) > 45% with histological evidence of iron overload
  * Alpha-1-antitrypsin (A1AT) phenotype/genotype ZZ or SZ
  * Wilson's disease
* Serum alanine aminotransferase (ALT) greater than 300 IU/L
* History of biliary diversion
* History of kidney disease and/or estimated glomerular filtration rate (eGFR) < than 60 mL/min/1.73 m2 using Schwartz Bedside GFR Calculator for Children isotope dilution mass spectroscopy (IDMS)-traceable
* Known Human Immunodeficiency Virus (HIV) infection
* Active, serious medical disease with life expectancy less than 5 years
* Active substance abuse including inhaled or injected drugs, in the year prior to screening
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding
* Participation in an investigational new drug (IND) trial in the 150 days prior to randomization
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* Inability to swallow capsules
* Known allergy to losartan potassium or other angiotensin receptor blocker
* Failure of parent or legal guardian to give informed consent or subject to give informed assent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Northwestern Univ-Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Results information from this trial will be submitted to ClinicalTrials.gov and a public use database deposited with the NIDDK Central Repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data from this study may be requested from the NIDDK Central Repository (https://www.niddkrepository.org/search/study/) two years after the completion of the primary outcome.
Access Criteria: Apply through the NIDDK Central Repository:
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: Nonalcoholic Steatohepatitis Clinical Research Network Centers — http://jhuccs1.us/nash/open/centers/centers.htm
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan: 100 mg losartan once per day
- Placebo: Matching placebo, taken once per day
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 43 | 40
Completed | 33 | 34
Not Completed | 10 | 6
Not completed — Trial stopped early | 5 | 2
Not completed — Clinic closed due to COVID-19 pandemic | 5 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (2) | 13 (2) | 13 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 33 | 34 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 33 | 66
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 28 | 25 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 8 | 17
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 115 (50) | 126 (61) | 120 (55)
Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 59 (26) | 70 (38) | 64 (33)
Alkaline phosphate [Mean (Standard Deviation); unit: U/L] | 192 (114) | 202 (99) | 197 (106)
y-Glutamyltransferase [Mean (Standard Deviation); unit: U/L] | 53 (44) | 51 (28) | 52 (37)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.6 (0.3) | 0.6 (0.3) | 0.6 (0.3)
Direct bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 159 (44) | 155 (31) | 157 (38)
High-density lipoprotein [Mean (Standard Deviation); unit: mg/uL] | 39 (7) | 41 (9) | 40 (8)
Low-density lipoprotein [Mean (Standard Deviation); unit: mg/uL] | 91 (40) | 92 (22) | 91 (32)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 158 (105) | 128 (58) | 143 (87)
Fasting serum glucose [Median (Inter-Quartile Range); unit: mg/dL] | 91 [84 to 100] | 87 [81 to 96] | 89 [82 to 97]
Insulin [Median (Inter-Quartile Range); unit: umol/mL] | 29 [18 to 42] | 38 [21 to 44] | 32 [21 to 44]
Homeostasis model assessment (HOMA) score of insulin resistance [Median (Inter-Quartile Range); unit: mg/dL x umol/mL/405] — Insulin Resistance Index (HOMA-IR) measures insulin resistance, calculated by fasting insulin (umol/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance
  mg/dL x umol/mL/405 | 6.5 [3.9 to 10.7] | 8.3 [4.0 to 10.2] | 7.1 [4.0 to 10.2]
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.4 (0.6) | 5.4 (0.3) | 5.4 (0.5)
Height [Mean (Standard Deviation); unit: cm] | 165 (9) | 165 (9) | 165 (9)
Weight [Mean (Standard Deviation); unit: kg] | 95 (17) | 96 (19) | 95 (18)
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 34 (5) | 35 (5) | 35 (5)
Mid arm circumference [Mean (Standard Deviation); unit: cm] | 33 (4) | 33 (4) | 33 (4)
Waist circumference [Median (Standard Deviation); unit: cm] | 108 (11) | 111 (11) | 110 (11)
Hip circumference [Median (Standard Deviation); unit: cm] | 110 (11) | 112 (11) | 111 (11)
Waist to hip ratio [Mean (Standard Deviation); unit: ratio] | 0.99 (0.06) | 0.99 (0.06) | 0.99 (0.06)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121 (9) | 119 (9) | 120 (9)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69 (6) | 69 (6) | 69 (6)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 79 (13) | 80 (13) | 79 (13)
Breath rate [Mean (Standard Deviation); unit: breaths/minute] | 18 (3) | 19 (4) | 19 (3)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.5 (1.1) | 14.0 (1.2) | 14.2 (1.2)
Hematocrit [Mean (Standard Deviation); unit: percentage of hematocrit] | 43.2 (3.3) | 42.0 (3.4) | 42.6 (3.4)
MCV [Mean (Standard Deviation); unit: fL] | 84.9 (4.4) | 84.7 (3.4) | 84.8 (4.0)
White blood cell count (WBC) [Mean (Standard Deviation); unit: 10^3 cells/uL] | 7.2 (1.5) | 8.6 (2.4) | 7.9 (2.1)
Red blood cell count (RBC) [Mean (Standard Deviation); unit: million cells/uL] | 509 (39) | 496 (37) | 503 (39)
Neutrophils [Mean (Standard Deviation); unit: cells/uL] | 3541 (1123) | 4231 (1867) | 3869 (1552)
Lymphocytes [Mean (Standard Deviation); unit: cells/uL] | 2656 (727) | 3031 (1003) | 2835 (884)
Monocytes [Median (Standard Deviation); unit: cells/uL] | 501 (165) | 578 (217) | 537 (194)
Eosinophils [Median (Standard Deviation); unit: cells/uL] | 297 (245) | 278 (249) | 288 (245)
Basophils [Mean (Standard Deviation); unit: cells/uL] | 35 (37) | 65 (126) | 49 (91)
Platelet [Median (Standard Deviation); unit: 1000 cells/mm^3] | 277 (57) | 311 (66) | 293 (64)
Sodium [Median (Standard Deviation); unit: mEq/L] | 140.0 (2.0) | 139.7 (2.0) | 139.9 (2.0)
Potassium [Median (Standard Deviation); unit: mEq/L] | 4.1 (0.3) | 4.2 (0.2) | 4.2 (0.3)
Chloride [Median (Standard Deviation); unit: mEq/L] | 103.9 (2.7) | 102.9 (2.5) | 103.4 (2.6)
Bicarbonate [Median (Standard Deviation); unit: mEq/L] | 24.3 (2.5) | 24.7 (2.0) | 24.4 (2.3)
Calcium [Median (Standard Deviation); unit: mEq/L] | 9.8 (0.4) | 9.8 (0.3) | 9.8 (0.3)
Blood urea nitrogen [Median (Standard Deviation); unit: mg/dL] | 10.9 (3.1) | 10.5 (2.5) | 10.7 (2.8)
Creatinine [Median (Standard Deviation); unit: mg/dL] | 0.56 (0.14) | 0.56 (0.13) | 0.56 (0.14)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 156 (19) | 155 (17) | 156 (18)
Prothrombin time [Mean (Standard Deviation); unit: seconds] | 12.3 (1.3) | 11.9 (1.3) | 12.1 (1.3)
International normalized ratio (INR) [Mean (Standard Deviation); unit: ratio] | 1.04 (0.07) | 1.04 (0.08) | 1.04 (0.07)
Uric acid [Median (Standard Deviation); unit: mg/dL] | 6.6 (1.7) | 6.6 (1.5) | 6.6 (1.6)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] | 3.8 (2.5) | 3.8 (3.0) | 3.8 (2.7)
Time from liver biopsy [Mean (Standard Deviation); unit: years] | 0.7 (0.6) | 0.8 (0.6) | 0.8 (0.6)
Nonalcoholic fatty liver disease (NAFLD) activity score [Mean (Standard Deviation); unit: units on a scale] — The Nonalcoholic fatty liver disease (NAFLD) Activity Score (NAS) is a composite score equal to the sum of the steatosis grade (0-3), lobular inflammation grade (0-3), and hepatocellular ballooning grade (0-2), from centralized pathologist scoring of liver biopsies. The overall scale of the NAS is 0-8, with higher scores indicating more severe disease.
  units on a scale | 4.6 (1.5) | 4.4 (1.2) | 4.5 (1.4)
Steatohepatitis Diagnosis [Count of Participants; unit: Participants] — Steatohepatitis diagnosis is based on central pathologists' review of liver biopsies. NAFLD, but not NASH was defined by at least 5% steatosis with or without inflammation but without ballooning injury. Borderline zone 3 pattern and borderline zone 1 pattern steatohepatitis had some but not all features of definite steatohepatitis, usually consisting of steatosis, inflammation, and fibrosis without ballooning. Definite steatohepatitis was defined by the presence of macrovesicular steatosis, inflammation, and hepatocellular ballooning. Definite steatohepatitis is considered a worse outcome.
  Participants
    NAFLD, not NASH | 15 | 9 | 24
    Borderline Zone 3 | 9 | 7 | 16
    Borderline Zone 1 | 11 | 12 | 23
    Definite steatohepatitis | 8 | 12 | 20
Fibrosis stage [Count of Participants; unit: Participants] — The amount of fibrosis is based on central pathologist grading of liver biopsies: 0=no fibrosis present; 1a=mild, zone 3 perisinusoidal fibrosis, 1b=moderate, zone 3, perisinusoidal fibrosis, 1c=portal/periportal fibrosis only, 2=zone 3 and periportal fibrosis, any combination, 3=bridging fibrosis. Fibrosis stages 1a, 1b, 1c recoded as 1, so the possible range of values for fibrosis stage was 0-3. Higher stage indicates worse outcome.
  Participants
    Stage 0 | 17 | 7 | 24
    Stage 1 | 13 | 20 | 33
    Stage 2 | 8 | 5 | 13
    Stage 3 | 5 | 8 | 13
Hepatocellular ballooning grade [Count of Participants; unit: Participants] — Hepatocellular ballooning grade based on pathologists' centralized scoring of liver biopsies. Hepatocellular ballooning grade scored as 0=none, 1=few ballooned hepatocytes, and 2=many ballooned hepatocytes. Higher values indicate worse outcome.
  Participants
    0 - None | 31 | 27 | 58
    1 - Few | 6 | 10 | 16
    2 - Many | 6 | 3 | 9
Steatosis [Count of Participants; unit: Participants] — Steatosis score is based on central pathologists' grading of liver biopsies: 0=<5% steatosis; 1=5-33% steatosis, 2=34-66% steatosis, 3=>66% steatosis. Higher values indicate worse outcome.
  Participants
    5-33% | 4 | 6 | 10
    34-66% | 13 | 11 | 24
    >66% | 26 | 23 | 49
Lobular inflammation [Count of Participants; unit: Participants] — The amount of lobular inflammation is based on central pathologists' grading of liver biopsies, and combines mononuclear, fat granulomas, and polymorphonuclear (pmn) foci: 0=none; 1=<2 under 20x magnification, 2=2-4 under 20x magnification, 3=>4 under 20x magnification. Lobular inflammation score has a possible range of 0 to 3. Higher values indicating a worse outcome.
  Participants
    <2 under 20x magnification | 21 | 17 | 38
    2-4 under 20x magnification | 16 | 21 | 37
    >4 under 20x magnification | 6 | 2 | 8
Portal inflammation [Count of Participants; unit: Participants] — The amount of portal inflammation is based on central pathologists' grading of liver biopsies: 0=none; 1=mild, 2=more than mild. Higher values indicate worse outcome.
  Participants
    None | 7 | 5 | 12
    Mild | 30 | 28 | 58
    More than mild | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Alanine Aminotransferase (ALT) From Baseline.
Description: Change ALT value in U/L (24 weeks minus baseline). A negative score indicates improvement.
Time Frame: Baseline and 24 weeks
Population: Results based on complete case analysis.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
U/L | -5.3 (51.4) | -6.3 (77.5)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = .95, ANCOVA; Adjusted for baseline value of ALT; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-30.6 to 32.7]

2. Secondary Outcome: Change in Gamma-glutamyl Transpeptidase (GGT) Compared to Baseline
Description: Change from baseline in gamma-glutamyl transpeptidase (GGT), measured in U/L.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
U/L | -1.9 (13.9) | 0.6 (19.7)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.56, ANCOVA; Adjusted for baseline value of GGT; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-11.0 to 6.0]

3. Secondary Outcome: Change in Serum Aspartate Aminotransferase AST at 24 Weeks Compared to Baseline AST
Description: Change from baseline in serum aspartate aminotransferase, measured in U/L.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
U/L | 0.2 (27.2) | -4.5 (37.0)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.53, ANCOVA; Adjusted for the baseline AST value; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-10.3 to 19.8]

4. Secondary Outcome: Relative Change in Serum Alanine Aminotransferase (ALT) Compared to Baseline ALT
Description: Relative change from baseline in serum ALT, measured in percentage of change.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
percentage of change | 2.7 (43.8) | -5.7 (73.2)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.57, ANCOVA; Adjusted for the baseline ALT value; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [-20.8 to 37.5]

5. Secondary Outcome: Change in ALT at 12 Weeks Compared to Baseline ALT
Description: Change from baseline in ALT at 12 weeks, measured in U/L.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL | -5.8 (43.0) | -19.3 (38.5)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority — Adjusted for the baseline ALT value; p = 0.25, ANCOVA; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [9.7 to 36.7]

6. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) Compared to Baseline.
Description: Homeostasis Model Assessment of Insulin Resistance Index (HOMA-IR) measures insulin resistance, calculated by fasting insulin (umol/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL x uU/mL/405
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL x uU/mL/405 | 4.5 (8.1) | 1.1 (5.2)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.05, ANCOVA; Adjusted for the baseline HOMA-IR value; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [0.0 to 6.8]

7. Secondary Outcome: Change in Weight at 24 Weeks Compared to Baseline
Description: Change from baseline in weight, measured in kg.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
kg | 4.4 (4.2) | 3.9 (4.3)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.64, ANCOVA; Adjusted for the baseline weight value; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.5]

8. Secondary Outcome: Change in Body Mass Index (BMI) at 24 Weeks Compared to Baseline.
Description: Change from baseline in BMI, measured in kg/m^2.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
kg/m^2 | 0.8 (1.2) | 0.8 (1.3)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.98, ANCOVA; Adjusted for the baseline BMI value; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.6]

9. Secondary Outcome: Change in Waist Circumference at 24 Weeks Compared to Baseline
Description: Change from baseline in waist circumference, measured in centimeters.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
cm | 2.6 (5.4) | 0.1 (6.4)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.10, ANCOVA; Adjusted for the baseline waist circumference value; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-0.5 to 5.3]

10. Secondary Outcome: Change in Waist-to-hip Ratio at 24 Weeks Compared to Baseline
Description: Change from baseline in waist-to-hip ratio, measured as the circumference of the waist in centimeters divided by the circumference of the hips in centimeters.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
ratio | 0.01 (0.05) | -0.01 (0.06)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.08, ANCOVA; Adjusted for the baseline waist-to-hip ratio; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0.00 to 0.05]

11. Secondary Outcome: Change in Pediatric Quality of Life Inventory (PedsQOL) Physical Health Score at 24 Weeks Compared to Baseline
Description: Pediatric Quality of Life Inventory (PedsQOL) version 4.0 is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Scores are transformed on a scale from 0 to 100, with higher scores indicating better health-related quality of life. Physical Health Summary Score =Physical Functioning Scale Score. The outcome is 24-week change from baseline in PedsQOL Physical Health Score, where higher values indicate improvement in quality of life.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
score on a scale | 0.9 (14.7) | -2.2 (13.3)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.29, ANCOVA; Adjusted for the baseline PedsQOL Physical Health score; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-2.8 to 9.0]

12. Secondary Outcome: Frequency of Adverse Events Over 24 Weeks
Description: Numbers of adverse events reported over 24 weeks.
Time Frame: Baseline and 24 weeks
Measure: Number; unit: adverse events
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
adverse events | 44 | 55
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.17, Exact conditional binomial test

13. Secondary Outcome: Change in Total Cholesterol at 24 Weeks Compared to Baseline
Description: Change from baseline in total cholesterol, measured in mg/dL
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL | -6.7 (28.4) | -4.1 (25.2)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.64, ANCOVA; Adjusted for baseline total cholesterol value; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-13.9 to 8.7]

14. Secondary Outcome: Change in Triglycerides at 24 Weeks Compared to Baseline
Description: Change from baseline in triglycerides, measured in mg/dL
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL | 13.2 (98.1) | 6.2 (41.1)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.67, ANCOVA; Adjusted for baseline triglyceride value; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [-25.6 to 39.7]

15. Secondary Outcome: Change in HDL Cholesterol at 24 Weeks Compared to Baseline
Description: Change from baseline in HDL cholesterol, measured in mg/dL
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL | -2.1 (6.2) | -1.1 (4.9)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.45, ANCOVA; Adjusted for baseline HDL cholesterol value; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.4 to 1.5]

16. Secondary Outcome: Change in LDL Cholesterol at 24 Weeks Compared to Baseline
Description: Change from baseline in LDL cholesterol, measured in mg/dL
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
mg/dL | -6.7 (29.2) | -6.2 (14.8)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.93, ANCOVA; Adjusted for baseline LDL cholesterol value; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-10.3 to 9.4]

17. Secondary Outcome: Change in Pediatric Quality of Life Inventory (PedsQOL) Psychosocial Health Score at 24 Weeks Compared to Baseline
Description: Pediatric Quality of Life Inventory (PedsQOL) version 4.0 is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Scores are transformed on a scale from 0 to 100, with higher scores indicating better health-related quality of life. Psychosocial Health Summary Score = Sum of items over the number of items answered in the Emotional, Social, and School Functioning Scales. The outcome is 24-week change from baseline in PedsQOL Psychosocial Health Score, where higher values indicate improvement in quality of life.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Losartan Potassium Capsule | Placebo Losartan Capsule
Number analyzed (Participants) | 33 | 34
score on a scale | 2.7 (12.2) | -0.2 (13.9)
Statistical Analysis 1: Comparison: Losartan Potassium Capsule vs Placebo Losartan Capsule; Test type: Superiority; p = 0.29, ANCOVA; Adjusted for baseline PedsQOL Psychosocial Health score; Median Difference (Final Values) = 2.9, 95% CI 2-sided [-2.5 to 20.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a time period of 36 weeks.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 4/40
Other Adverse Events (participants affected / at risk) | 28/43 | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=43) | Placebo (N=40)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Surgical and medication procedures - Other, bilateral knee surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Bilateral knee surgery for genu valgum
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=43) | Placebo (N=40)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 7 (7)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder, other - knee injury, pain, bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder, other-slipped capital femoral epiphysis (SCFE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Rhinoseptoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Rash, pustular (Infections and infestations) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitus (Infections and infestations) | 2 (2) | 1 (1)
Sore throat (Infections and infestations) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
Viremia (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03467217/Prot_SAP_000.pdf
  • Informed Consent Form: Parental Permission Form (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03467217/ICF_001.pdf
  • Informed Consent Form: Child Assent Form (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03467217/ICF_002.pdf
  • Informed Consent Form: HIPAA Authorization Form (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03467217/ICF_003.pdf